CLINICAL TRIAL: NCT06741969
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Phase 3 Protocol to Assess the Efficacy and Safety of Nipocalimab in Adults With Moderate to Severe Sjogren's Disease (SjD)
Brief Title: Nipocalimab in Moderate to Severe Sjogren's Disease
Acronym: DAFFODIL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 80202135SJS3001; 80202135SJS3001 (Other: Janssen Research & Development, LLC); 2024-513965-38-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-12-18; First posted 2024-12-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Sjogrens Syndrome
Keywords: Sjogrens Disease
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 2 identical studies (conducted under this single protocol) to make a total of 300 participants in each study. Participants in each study will be randomly assigned to one of the arms nipocalimab or placebo respectively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nipocalimab (Experimental): Participants will receive nipocalimab subcutaneously (SC) along with standard of care treatments. At the Week 48 visit, eligible participants from both studies will have the option to enter an open-label long-term extension (OLE) phase, where they will continue to receive nipocalimab until Week 143 or until the study intervention is discontinued and participants opt to withdraw from the study.
  Interventions: Drug: Nipocalimab; Drug: Standard of care treatment
- Placebo (Placebo Comparator): Participants will receive placebo subcutaneously along with standard of care treatments. At the Week 48 visit, eligible participants from both studies will have the option to enter an OLE phase, where they will receive nipocalimab until Week 143 or until the study intervention is discontinued and participants opt to withdraw from the study.
  Interventions: Drug: Placebo; Drug: Standard of care treatment

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab SC.
  Other Names: JNJ-80202135, JNJ-86507083, M281
  Arms: Nipocalimab
Drug: Placebo — Placebo SC.
  Arms: Placebo
Drug: Standard of care treatment — Protocol-defined topical and systemic standard of care background treatments.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of nipocalimab in participants with moderate to severe Sjogren's disease (SjD).

DETAILED DESCRIPTION:
This clinical development program for nipocalimab in SjD includes 2 identical double blind, placebo-controlled studies to evaluate the efficacy, safety, and tolerability of nipocalimab in participants greater than or equal to (>=) 18 years of age with moderate to severe SjD.

ELIGIBILITY:
Inclusion Criteria:-

* Medically stable on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and 12-lead electrocardiogram (ECG) performed at screening
* Meets criteria for diagnosis of SjD by the 2016 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) classification criteria
* Seropositive for antibodies to Ro/SSA (Ro60 and/or Ro52) at screening
* Total ClinESSDAI score greater than or equal to (>=) 5 at screening
* Participants of childbearing potential must have a negative highly sensitive serum (beta-hCG) pregnancy test at screening and a negative urine pregnancy test at Week 0 prior to randomization

Exclusion Criteria:

* Has a history of severe, progressive and/or uncontrolled hepatic, gastrointestinal, renal, pulmonary, cardiovascular, psychiatric, neurological or musculoskeletal disorder, hypertension, and/or any other medical or uncontrolled autoimmune disorder or clinically significant abnormalities in screening laboratory
* Known allergies, hypersensitivity, or intolerance to nipocalimab or its excipients or excipients used in the placebo formulation
* Has any confirmed or suspected clinical immunodeficiency syndrome not related to treatment of his/her SjD or has a family history of congenital or hereditary immunodeficiency
* Has shown a previous severe immediate hypersensitivity reaction, such as anaphylaxis, to therapeutic proteins (for example [e.g.], monoclonal antibodies, intravenous immunoglobulin)
* Has any unstable or progressive manifestation of SjD that is likely to warrant escalation in therapy beyond permitted background medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-08-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (ClinESSDAI) Score at Week 48 | Baseline to Week 48
  ClinESSDAI is a validated tool used in clinical studies to measure the systemic disease activity in participants with SjD. The ClinESSDAI includes 11 domains divided into 3-4 activity levels, where zero represents no activity and low, medium, and high scores can vary in numerical value depending on the domain being measured. A higher score represents worse disease symptoms.

SECONDARY OUTCOMES:
Improvement from Baseline in Minimal Clinically Important Improvement (MCII) in ClinESSDAI Score at Week 48 | Baseline to Week 48
  The ClinESSDAI is a validated tool used in clinical studies to measure the systemic disease activity in participants with Sjogren's syndrome.
Improvement from Baseline in ClinESSDAI Score at Week 48 in Participants with High Immunoglobulin (IgG) Levels at Baseline | Baseline to Week 48
  ClinESSDAI is a validated tool used in clinical studies to measure the systemic disease activity in participants with SjD.
Change from Baseline in ClinESSDAI Score at Week 8 | Baseline to Week 8
  ClinESSDAI is a validated tool used in clinical studies to measure the systemic disease activity in participants with SjD.
Change from Baseline in Stimulated Salivary Flow Rate at Week 48 | Baseline to Week 48
  Stimulated salivary flow is considered a reliable and objective method to evaluate glandular function in SjD patients.
Change from Baseline in Sjogren's Symptoms Dryness Score at Week 48 | Baseline to Week 48
  Participants will be asked to report the worst severity of their dryness symptoms on a 0 to 10 numeric rating scale (NRS), with score 0 indicating "No [specific symptom]" and score 10 indicating "Severe [specific symptom]". Higher scores reflect greater symptom severity. Change from baseline in Sjogren's Symptoms dryness score at Week 48 for US, US reference regions, and other non-US regions will be reported.
Change from Baseline in Sjogren's Symptoms Joint Pain Score at Week 48 | Baseline to Week 48
  Participants will be asked to report the worst severity of their joint pain symptoms on a 0 to 10 numeric rating scale (NRS), with score 0 indicating "No [specific symptom]" and score 10 indicating "Severe [specific symptom]". Higher scores reflect greater symptom severity. Change from baseline in Sjogren's Symptoms joint pain score at Week 48 for US, US reference regions, and other non-US regions will be reported.
Change from Baseline in EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) Score At Week 48 | Baseline to Week 48
  ESSPRI is a participant-reported assessment of the severity of dryness, fatigue, and pain associated with primary Sjogren's Syndrome. Participants are asked to rate the severity of dryness, fatigue, and pain on a 0 to 10 NRS, with score 0 indicating "No [specific symptom]" and score 10 indicating "Severe [specific symptom]". A global score, calculated as the mean of the 3 domain scores, ranges from 0 to 10, with higher scores reflecting greater (worse) symptom severity. Change from baseline in Sjogren's Symptoms score at Week 48 for EU, UK & EU reference regions will be reported.
Change from Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT) Fatigue Score at Week 48 | Baseline to Week 48
  FACIT-Fatigue version 4.0 is a 13-item questionnaire that assesses participant-reported fatigue and its impact upon daily activities and function over the past 7 days. Participants will be asked to answer each question using a 5-point Likert scale (0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; and 4=Very much). FACIT-Fatigue has a total score range from 0 to 52, with 0 being the worst possible score and 52 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (245):
- United States (43):
  - Advanced Clinical Research Center, Chula Vista, California
  - Providence Medical Foundation, Fullerton, California
  - Arthritis & Osteoporosis Medical Center - La Palma, La Palma, California
  - NovaMed Research, Monterey Park, California
  - Medvin Clinical Research San Leandro, San Leandro, California
  - Providence Saint John s Health Center, Santa Monica, California
  - Solace Clinical Research California, Tustin, California
  - Inland Rheumatology Clinical Trials Inc., Upland, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Clinical Research of West Florida Inc, Clearwater, Florida
  - UF Health Rheumatology, Jacksonville, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Sarasota Arthritis Center, Sarasota, Florida
  - BioResearch Partner, South Miami, Florida
  - Immunology and Rheumatology Research Associates LLC, Suwanee, Georgia
  - Clinical Investigation Specialists - Clinic of Robert Hozman, Skokie, Illinois
  - Willow Rheumatology and Wellness PLLC, Willowbrook, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - St. Paul Rheumatology P A, Eagan, Minnesota
  - AARA Clinical Research- Kansas City Physicians Partners, Kansas City, Missouri
  - Arthritis Rheumatic And Back Disease Associates, Voorhees Township, New Jersey
  - NYU Langone Health - Clinical and Translational Science Institute, New York, New York
  - Pioneer Clinical Research NY, New York, New York
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Atrium Health SouthPark Rheumatology, Charlotte, North Carolina
  - Onsite Clinical Solutions, Salisbury, North Carolina
  - Wright State Physicians Health Center, Fairborn, Ohio
  - OMRF Rheumatology Center of Excellence, Oklahoma City, Oklahoma
  - Rheumatology Associates of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Philadelphia, Philadelphia, Pennsylvania
  - Low Country Rheumatology PA, Summerville, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - AARA Clinical Research - Murfreesboro Medical Clinic, Murfreesboro, Tennessee
  - Amarillo Premier Research, Amarillo, Texas
  - Texas Rheumatology Research Institute LLC, Plano, Texas
  - Fort Bend Rheumatology Associates PLLC, Sugar Land, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - Alpine Research TC LLC, Layton, Utah
  - Tidewater Clinical Research, Chesapeake, Virginia
  - Overlake Arthritis and Osteoporosis Center, Bellevue, Washington
- Argentina (10):
  - Instituto Medico De Alta Complejidad (IMAC), Buenos Aires
  - Centro de Investigacion San Miguel CISM, Buenos Aires
  - Mautalen Salud e Investigacion, CABA
  - Centro Medico del Dr. Javier Gerardo Tartaglione, Cdad Autonoma de Buenos Aires
  - Centro de Investigacion en Enfermedades Reumaticas CIER, Ciudad de Buenos Aires
  - Centro Medico Barrio Parque. Swiss Medical Group, Ciudad de Buenos Aires
  - Cosultorios Reumatologógicos Pampa, Ciudad de Buenos Aires
  - Cer Instituto Medico, Quilmes
  - MR Medicina Reumatologica, San Fernando
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Austria (5):
  - Medizinische Universitaet Graz, Graz
  - SCRI CCCIT gem GmbH, Salzburg
  - LK Weinviertel Stockerau, Stockerau
  - Medizinische Universitaet Wien, Vienna
  - Wiener Gesundheitsverbund Klinik Hietzing, Vienna
- Brazil (13):
  - Instituto D Or de Pesquisa e Ensino, Brasília
  - Ceti - Centro de Estudos Em Terapias Inovadoras, Curitiba
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - LMK Servicos Medicos S S, Porto Alegre
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto, Ribeirão Preto
  - SER - Servicos Especializados em Reumatologia da Bahia, Salvador
  - Instituto D Or de Pesquisa e Ensino, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - EBSERH Empresa de Servicos Hospitalares Hospital Samaritano, São Paulo
  - CEPIC Centro Paulista de Investigacao Clinica e Servicos Medicos, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
  - CEDOES Centro de Pesquisa Clinica e Diagnostico do Espirito Santo Ltda, Vitória
- Bulgaria (9):
  - UMHAT Kaspela, Plovdiv
  - Medical Center Artmed, Plovdiv
  - Medical Center Teodora, Rousse
  - Lyulin Multi Profile Hospital For Active Medical Treatment, Sofia
  - Diagnostic-Consultative Center (DCC) Aleksandrovska, Sofia
  - St Ivan Rilski University Multiprofile Hospital For Active Treatment, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Diagnostic Consultative Center - DCC Equita EOOD, Varna
  - MHAT 'St. Marina' EAD, Varna
- Canada (3):
  - Dr Sabeen Anwar Medicine Professional Corporation, Windsor, Ontario
  - Hospital Regional de Rimouski, Rimouski, Quebec
  - Centre de Recherche Musculo Squelettique, Trois-Rivières, Quebec
- China (30):
  - Beiijing Friendship Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - Dazhou Central Hospital, Dazhou
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Shandong Provincial Hospital, Jinan
  - Jinhua municipal central hospital, Jinhua
  - Linyi City People Hospital, Linyi
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Zhongda Hospital Southeast University, Nanjing
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Ningbo medical center lihuili hospital, Ningbo
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - Shenshan Medical Center Memorial Hospital of Sun Yat Sen University, Shanwei
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Academy of Medical Sciences, Taiyuan
  - Tianjin First Central Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The first affiliated hospital of xiamen university, Xiamen
  - Xinxiang Central Hospital, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - People s Hospital of Ningxia Hui Autonomous Region, Yinchuan
  - Zhongshan Traditional Chinese Medicine Hospital, Zhongshan
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Zealand University Hospital, Køge
- France (8):
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - CHU Dijon Bourgogne - Hopital Francois Mitterrand, Dijon
  - Hopital Bicetre Aphp Hopitaux Universitaires Paris Sud, Le Kremlin-Bicêtre
  - CHRU de Lille Hopital Claude Huriez, Lille
  - CHRU Montpellier Hopital Lapeyronie, Montpellier
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHRU de Strasbourg - Hopital de Hautepierre, Strasbourg
  - CHU Bordeaux, Talence
- Germany (11):
  - Krankenhaus Porz am Rhein, Cologne
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Erlangen Medizinische Klinik 3, Erlangen
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Rheumazentrum Ruhrgebiet, Herne
  - Klinikum der Universitaet Muenchen, München
  - Medicover Muenchen Ost MVZ, München
  - Rheumazentrum Ratingen, Ratingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hungary (7):
  - Semmelweis Egyetem Reumatologiai es Immunologiai Klinika, Budapest
  - Betegapolo Irgalmas Rend Budai Irgalmasrendi Korhaz, Budapest
  - Clinexpert Kft, Budapest
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szegedi Tudomanyegyetem, Szeged
  - Vita Verum Medical Egeszsegugyi Szolgaltato Bt, Székesfehérvár
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Tzafon Medical Center Poria, Har Poriyya
  - Galil Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Ospedale San Raffaele, Milan
  - Centro Specialistico Ortopedico Traumatologico Gaetano Pini CTO, Milan
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera di Perugia Ospedale S.Maria della Misericordia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Umberto I Policlinico di Roma, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Campus Bio Medico di Roma, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale S. Maria Della Misericordia, Udine
- Japan (12):
  - St. Luke's International Hospital, Chūōku
  - Tokyo Metropolitan Tama Medical Center, Fuchū
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Shinkenko Clinic, Naha
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Hokkaido University Hospital, Sapporo
  - Sasebo Chuo Hospital, Sasebo
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga Gun
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - Nihon University Itabashi Hospital, Tokyo
- Mexico (8):
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa, Culiacán
  - Clinica de Investigacion en Reumatologia y Obesidad, Guadalajara
  - Centro Medico Nacional Siglo XXI IMSS, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico D F
  - Medical Care & Research SA de CV, Mérida
  - CITER Centro de Investigacion y Tratamiento de las Enfermedades Reumaticas S A de C V, México
  - SMIQ S de R L de C V, Querétaro
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi, San Luis Potosí City
- Poland (14):
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - ETG Debica, Dębica
  - Malopolskie Badania Kliniczne Sp z o o, Krakow
  - Futuremeds Krakow, Krakow
  - ETG Lublin Poradnie Specjalistyczne, Lublin
  - Etyka Osrodek Badan Klinicznych Tomasz Pesta S K A, Olsztyn
  - AI Centrum Medyczne, Poznan
  - ETG Siedlce, Siedlce
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
  - FutureMeds Targowek, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - FutureMeds Wroclaw, Wroclaw
- Portugal (4):
  - Ipr Inst Port de Reumatologia, Lisbon
  - Uls Lisboa Ocidental - Hosp. Egas Moniz, Lisbon
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Uls Gaia Espinho, Vila Nova de Gaia
- Romania (7):
  - Spitalul Clinic Sf Maria, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Policlinica CCBR SRL, Bucharest
  - Hiperdia SA, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Medisof Diagnostic S R L, Craiova
  - Selfmed Clinique S.R.L., Timișoara
- South Korea (8):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - The Catholic university of Korea, St. Vincent's Hospital, Suwon
  - Ajou University Hospital, Suwon
- Spain (8):
  - Hosp. Cima Sanitas Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Gral. Juan Ramon Jimenez, Huelva
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. de Navarra, Pamplona
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Infanta Luisa, Seville
- Universitatsspital Basel, Basel, Switzerland
- Taiwan (7):
  - NTU Biomedical Park Hospital, Hsinchu
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (6):
  - Gulhane Training and Research Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Uludag University Medical Faculty, Bursa
  - Marmara University Istanbul Pendik Education and Research Hospital, Istanbul
  - Necmettin Erbakan University, Konya
- United Kingdom (8):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Doncaster Royal Infirmary, Doncaster
  - Barts Health NHS Trust, Greater London
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospital Aintree, Liverpool
  - West Middlesex University Hospital, London
  - Peterborough City Hospital, Peterborough
  - Great Western Hospital, Swindon

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency